CLINICAL TRIAL: NCT01823770
Title: Effect of Rotigotine Patch Treatment on Cardiovascular Markers in Idiopathic Restless Legs Syndrome : a Pilot Randomized, Placebo-controlled Study
Brief Title: Effect of Rotigotine Patch Treatment on Cardiovascular Markers in Idiopathic Restless Legs Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8917
Record Dates: First submitted 2013-03-22; First posted 2013-04-04 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Restless Legs Syndrome (RLS)
Keywords: Restless Legs Syndrome (RLS); Rotigotine; HTA; Cardiovascular diseases; Periodic Limb Movements in Sleep (PLMS); dopaminergic agonist; Sympathetic overactivity; blood pressure
MeSH Terms: conditions — Restless Legs Syndrome; Cardiovascular Diseases | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rotigotine (Active Comparator): Patients randomized to rotigotine who will be treated with rotigotine patchs
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Patients randomized on the placebo group who will be treated with placebo patchs
  Interventions: Drug: Placebo patchs
- Control group (No Intervention): Volunteers matched on sex, age and BMI with RLS patients who will not receive treatment(no treatment)

INTERVENTIONS:
Drug: Rotigotine — Subjects randomized to rotigotine will start treatment with a rotigotine dose of 1mg/24h for 1 week. The dose can be increased weekly until either the optimal or the maximal dose of 3mg/24h has been reached. Subjects will maintain the optimal/maximal dose during the 2-week Maintenance Period. Following the Maintenance Period, subjects will be de-escalated from their optimal dose by decreasing the dose by 1mg/24h every other day until complete withdrawal (Taper period).
  Other Names: Rotigotine patchs
  Arms: Rotigotine
Drug: Placebo patchs — Subject randomized on the placebo group will be treated with placebo patchs, following the same modalities and study periods that the rotigotine arm
  Arms: Placebo

SUMMARY:
Several studies report association between restless legs syndrome (RLS), HTA and cardiovascular diseases .

The mechanisms involved in this relationship remained unknown, but several evidences favor the role of periodic limb movements in sleep (PLMS), patterns frequently associated with RLS. Sympathetic overactivity is associated with PLMS with increased pulse rate and blood pressure coincident with PLMS. PLMS-related repetitive nocturnal blood pressure fluctuations could contribute to the risk of high blood pressure, heart disease, and stroke in patients with RLS, especially in the elderly. Several studies already reported that dopaminergic agonists reduce the severity of RLS and the PLMS index.

Do dopaminergic agonists reduce the risk of cardiovascular diseases and associated autonomic dysfunctions in patients with RLS ?

Nocturnal BP (blood pressure) decline has major clinical implications, and the loss of normal reduction in BP during sleep is associated with high risk of cardiovascular morbidity and mortality.

The main aim of this study was to evaluate the impact of rotigotine patch treatment on validated cardiovascular risk factors ambulatory BP during night, day and night-to-day ratio, and endothelial function in patients with idiopathic RLS compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, all of the following criteria must be present in the patients:

  1. Subject is informed and given ample time and opportunity to think about her/his participation and has given her/his written informed consent.
  2. Subject understands the investigational nature of the study and is willing and able to comply with the study requirements. Subject is willing to accept that he/she might be treated with placebo during the Treatment Period.
  3. Subject is able to apply/remove the study patches correctly.
  4. Subject is male or female, and is ≥18 and ≤80 years of age.
  5. Subject has a body mass index (BMI) of ≥18kg/m2 and ≤35kg/m2.
  6. Subject has ferritin concentration of ≥50ng/mL at Screening.

  9. Subject has a diagnosis of RLS based on the 4 cardinal diagnostic clinical features according to the International Restless Legs Syndrome Study Group 11. At Baseline, subject has a score of ≥15 points on the IRLS (indicating moderateto severe RLS).

  12. At Baseline, subject scores ≥10 PLMs per hour on the PLMI based on PSG
* To be eligible to participate in this study, all of the following criteria must be present in the controls:

  1. Subject is informed and given ample time and opportunity to think about her/his participation and has given her/his written informed consent.
  2. Subject understands the investigational nature of the study and is willing and able to comply with the study requirements.

  4. Subject is male or female, and is ≥18 and ≤80 years of age. 5. Subject has a body mass index (BMI) of ≥18kg/m2 and ≤35kg/m2.

Exclusion Criteria:

* RLS patients are not permitted to be included in the study if any of the following criteria is met:

  1. Subject has RLS associated with previous or concomitant therapy with dopamine D2 receptor antagonists, butyrophenones, metoclopramide, atypical antipsychotics (eg, olanzapine), antidepressants, mianserine, or lithium or H2-blockers (eg, cimetidine).
  2. Subject has a history of any sleep disorder other than RLS including a severe obstructive sleep apnea syndrome (Apnea hypopnea index > 30/h) not treated by a controlled Continuous Positive Airway Therapy (CPAP) for at least 1 month prior to Screening, or has narcolepsy or other hypersomnia.
  3. Subject has clinically relevant polyneuropathy which cannot be clearly differentiated from RLS symptoms in the opinion of the investigator.
  4. Subject has additional clinically relevant concomitant diseases, such as attention deficit hyperactivity disorder, painful legs, and moving toes.
  5. Subject has other central nervous system diseases, such as Parkinson's disease, dementia, progressive supranuclear paresis, multisystem atrophy, Huntington's chorea, amyotrophic lateral sclerosis, or Alzheimer's disease.
  6. Subject has evidence of an impulse control disorder (Visit 1) as assessed by the Minnesota Impulsive Disorders Interview. If a subject has 1 or more positive modules on the mMIDI, he/she must be referred for a structured clinical interview, such as the Structured Clinical Interview for DSM-IV Axis 2 Personality Disorders (SCID-II) or another applicable structured interview for the diagnosis of ICDs.
  7. Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months.
  8. Subject has a prior history of psychotic episodes.
  9. Subject has a history of chronic alcohol or drug abuse within the prior 12 months.
  10. Subject has any medical or psychiatric condition which in the opinion of the investigator, can jeopardize or compromise the subject's wellbeing or ability to participate in this study.
  11. Subject has a history of symptomatic (not asymptomatic) orthostatic hypotension in the 6 months prior to Baseline
  12. Subject has clinically relevant cardiovascular disease which, in the opinion of the investigator, can compromise the subject's wellbeing or ability to participate in this study.
  13. Subject has clinically relevant venous or arterial peripheral vascular disease.
  14. Subject has a malignant neoplastic disease requiring therapy within 12 months prior to Screening (Visit 1).
  15. Subject is currently receiving treatment with any of the following drug classes: neuroleptics, hypnotics, antidepressants, anxiolytic drugs, anticonvulsive therapy, budipine, dopamine antagonist antiemetics (except domperidone), opioids, benzodiazepines (zolpidem and zopiclone may be considered as rescue medication in case of inability to sleep), monoamine oxidase (MAO) inhibitors, catechol-O-methyltransferase (COMT) inhibitors, sedative antihistamines, psychostimulants, or amphetamines. If subject has received such therapy, a Washout Period of at least 7 days prior to Baseline is required before starting treatment in this study.
  16. Subject is pregnant, nursing, or is a woman of childbearing potential who is not surgically sterile, 2 years postmenopausal, or does not consistently use 2 combined effective methods of contraception (including at least 1 barrier method), unless sexually abstinent.
  17. Subject pursues shift work or performs other continuous non-disease-related life conditions which do not allow regular sleep at night.
  18. Subject has had previous treatment with dopamine agonists within a period of 14 days prior to Baseline, or L-dopa within 7 days prior to Baseline.
  19. Subject has a medical history indicating intolerability to dopaminergic therapy (if pretreated) or has experienced augmentation when previously treated with any dopaminergic agent.
  20. Subject has participated in another study of an investigational drug within the 28 days prior to Baseline or is currently participating in another study of an investigational drug.
  21. Subject has a known hypersensitivity to any of the components of the study medication, such as a history of significant skin hypersensitivity to adhesives, known hypersensitivity to other transdermal medications, or has unresolved contact dermatitis.
  22. Subjects unable or unwilling to undergo informed consent
  23. Subject with no rights from the national health insurance programme
  24. Subject has a medical history indicating intolerability to rotigotine or inefficiency (previously treated).
  25. subjects who is performed an IRM examen during the study duration.
* Normal controls are not permitted to enroll in the study if any of the following criteria is present:

  1. Subject has a diagnosis of RLS based on the 4 cardinal diagnostic clinical features according to the International Restless Legs Syndrome Study Group
  2. At Baseline, subject scores ≥10 PLMs per hour on the PLM index based on PSG
  3. Subject has a history of any sleep disorder including a severe obstructive sleep apnea syndrome (Apnea hypopnea index > 30/h) not treated by a controlled Continuous Positive Airway Therapy (CPAP) for at least 1 month prior to Screening, or has narcolepsy or other hypersomnia.
  4. Subject has clinically relevant polyneuropathy, attention deficit hyperactivity disorder, Parkinsonian syndrome or dementia
  5. Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months, or history of psychotic episodes, or history of chronic alcohol or drug abuse within the prior 12 months.
  6. Subject has clinically relevant cardiovascular disease which, in the opinion of the investigator, can compromise the subject's wellbeing or ability to participate in this study.
  7. Subject is currently receiving treatment with any of the following drug classes: dopaminergic agonists, neuroleptics, hypnotics, antidepressants, anxiolytic drugs, anticonvulsive therapy, budipine, dopamine antagonist antiemetics (except domperidone), opioids, benzodiazepines (zolpidem and zopiclone may be considered as rescue medication in case of inability to sleep), monoamine oxidase (MAO) inhibitors, catechol-O-methyltransferase (COMT) inhibitors, sedative antihistamines, psychostimulants, or amphetamines.
  8. Subject is pregnant, nursing, or is a woman of childbearing potential who is not surgically sterile, 2 years postmenopausal, or does not consistently use 2 combined effective methods of contraception (including at least 1 barrier method), unless sexually abstinent.
  9. Subject pursues shift work or performs other continuous non-disease-related life conditions which do not allow regular sleep at night.
  10. Subject has participated in another study of an investigational drug within the 28 days prior to Baseline or is currently participating in another study of an investigational drug
  11. Subjects unable or unwilling to undergo informed consent
  12. Subject with no rights from the national health insurance programme

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-11-26 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Percentages of non-dippers(defined as <10% drop in BP during sleep)at 35+/-3 days | 35 +/- 3 day
  Percentages of non-dippers is defined as <10% drop in blood pressure (BP) during sleep (24h ambulatory BP monitoring).

SECONDARY OUTCOMES:
Digital pulse amplitude measured by reactive hyperhemia with finger plethysmographic methodology | day 35 +/- 3
  Fasting morning peripheral arterial tonometry (PAT)
PLMS and PLMS-microarousal indexes | day 35 +/- 3
  Nocturnal polysomnography (PSG)
Amplitude of PLMS-related HR responses | day 35 +/- 3
  Nocturnal polysomnography (PSG)

OTHER OUTCOMES:
change from baseline score of International RLS severity scale ((IRLS), RLSQoL, CGI)) at 35+/-3 days | V0(Day -10± 3V1 (Day 0±3), V2(Day 14±3), V3(Day 21±3), V4(Day 35± 3)
  Questionnaires on Epworth, IRLSQ, RLS QoL, CGI
change from baseline "total sleep time" at 35 +/-3 days | At the first visit (day 0) and the forth visit (day 35 +/- 3)
  Nocturnal polysomnography (PSG)
change from baseline cytokine level at 35+/-3days | At the first visit (day 0) and the forth visit (day 35 +/- 3)
  Fasting morning blood sample
change from baseline % sleep stage at 35+/-3 days | At the first visit (day 0) and the forth visit (day 35 +/- 3)
  Nocturnal polysomnography (PSG)
change from baseline Lipid level at 35+/-3 days | At the first visit (day 0) and the forth visit (day 35 +/- 3)
  Fasting morning blood sample
change from baseline glucid level at 35+/-3days | At the first visit (day 0) and the forth visit (day 35 +/- 3)
  Fasting morning blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Yves Dauvilliers, PU PH, Principal Investigator — UH Montpellier
Locations (1):
- UH Montpellier, Montpellier, France